CLINICAL TRIAL: NCT06139783
Title: Combined Program of Supervised Physical Exercise and Nutritional Counseling in Ovarian Cancer Patients on Frontline Maintenance Treatment With PARP Inhibitors: ACTIVA Study
Brief Title: Combined Program of Supervised Physical Exercise and Nutritional Counseling in Ovarian Cancer Patients on Frontline Maintenance Treatment With PARP Inhibitors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncare Madrid (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACTIVA
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physycal Exercise (Experimental): Patients included in the study will follow an online physical exercise program supervised by a physical exercise specialist in which they will perform up to 300 minutes of moderate-intensity aerobic exercise or up to 150 minutes of vigorous aerobic exercise and 2 strength sessions per week for 12 weeks (following WHO recommendations for cancer survivors).
  Interventions: Procedure: Exercise and dietary recommendations

INTERVENTIONS:
Procedure: Exercise and dietary recommendations — Online physical exercise program and online nutritional assessment with personalized health and dietary recommendations

SUMMARY:
Patients will be recruited in the 4 participating sites and will sign the informed consent If they agree to participate. It is planned to include 32 patients with ovarian cancer on maintenance PARPi after response to first-line platinum-based chemotherapy in the study.

Patients included in the study will follow an online physical exercise program supervised by a physical exercise specialist in which they will perform up to 300 minutes of moderate-intensity aerobic exercise or up to 150 minutes of vigorous aerobic exercise and 2 strength sessions per week for 12 weeks (following World Health Organization (WHO) recommendations for cancer survivors).

DETAILED DESCRIPTION:
In an initial nursing visit, patient's demographic data, epidemiological, clinical, biological and training-related variables, as well as fatigue, quality of life and mental health questionnaires will be obtained. The activity bracelet, blood pressure monitor, elastic bands set, and a document of exercise compliance will also be provided to the patient. If necessary, a local gym registration will be provided.

The program will include 12 stages. Each stage will correspond to one week, with 3 to 5 sessions per week containing cardiorespiratory, strength and flexibility training tasks. Where necessary, joint mobility and neuromotor work will be included. The exercise prescription parameters will be adapted to the patient's clinical history (intensity, frequency, duration, training system, progression) and patient's interest if the clinical condition allows it. Throughout the program, periodic records of symptoms, effort and intensity scales, blood pressure, heart rate, as well as the patient's emotional state will be requested.

After the registration process, a tutor (physiotherapist) will be assigned to the patient. An initial assessment is scheduled to analyze the clinical situation and to design the program. During this first consultation, the patient will be introduced to the platform and will take a preliminary course on basic training for control and monitoring of the program.

During the course, questions can be asked to the tutor via the platform chat. Once the patient reports the completion of a stage, the subsequent content will be released.

The tutor will supervise and follow up through scheduled video calls (one every 15 days of training); as well as through the message system.

All patients will have a period of 12 weeks to complete their program. The tutor will maintain constant communication with the responsible physician.

Participants will also receive an initial and mid-program online nutritional assessment with personalized health and dietary recommendations.

A final nurse visit will be made at the end of the program and after 3 months of follow up to evaluate whether the patient maintains the healthy habits acquired during the 12 weeks of the program.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years old.
2. High grade serous or endometrioid ovarian, primary peritoneal or fallopian tube cancer.
3. Provide written informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Stage III-IV according to International Federation of Gynecology and Obstetrics (FIGO) staging system.
6. Life expectancy of ≥ 6 months.
7. Maintenance treatment with PARPi after response to first-line platinum-based chemotherapy, initiated at least 4 weeks prior to the informed consent signature.
8. Patient is clinically stable and anticipate remaining on therapy for the duration of the exercise program.
9. Patient is willing to provide a tumor tissue sample either collected from a prior biopsy or cytoreductive/debulking surgery occurring at any time since diagnosis, if available.
10. Patients with sufficient digital capacity at the investigator's discretion.
11. Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures.
12. Have adequate baseline function within 28 days of enrollment:

    * Platelets ≥ 100 × 109/L
    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Hemoglobin ≥ 9 g/dL or 5.6 mmol/L
    * Aspartate transaminase and alanine transaminase ≤2.5 × upper limit of normal (ULN), <5 × ULN in patients with known liver metastases
    * Serum total bilirubin ≤ 1.5 × ULN

      * 1.5-3.0 × ULN may be included with appropriate starting dose adjustment to 200 mg niraparib daily.
    * Creatinine <1.5 × ULN or estimated glomerular filtration rate (GFR) ≥50 ml/min by Cockcroft-Gault.

Exclusion Criteria:

1. Women with diagnosis of recurrent ovarian cancer.
2. Serous, non-healing wound, ulcer or bone fracture.
3. Active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder or coagulopathy.
4. Central nervous system disease.
5. History of significant cardiovascular disease within 6 months prior to enrollment:

   * History of NCI CTCAE v5.0 Grade ≥ 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) Class ≥ II.
   * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate ≥100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block, such as second-degree AV-block Type 2 [Mobitz II] or third-degree AV-block).
   * Myocardial infarction or ischemic disease,
   * Clinically significant valvular heart disease.
   * Ischemic or hemorrhagic stroke,
   * Thromboembolic events,
   * Peripheral vascular disease,
   * Aortic aneurysm, aortic dissection.
6. Pre-existing uncontrolled hypertension as documented by two baseline blood pressure readings taken at least five minutes apart, defined as systolic BP ≥ 140 or diastolic BP ≥ 90 mm Hg pressure.
7. Patient requires recurrent (≥ 1 per month) fluid drainage (eg, paracentesis, thoracocentesis, pericardiocentesis) or patient requires fluid drainage of ≥ 500 mL within 4 weeks of the expected date of exercise initiation.
8. Active infection and/or fever ≥ 38,5ºC within 7 days prior to initiation of the program requiring systemic antibiotics (excluding uncomplicated urinary tract infection).
9. Patient has undergone any major surgical procedure within 3 weeks prior to screening or is planned during the program.
10. Known QT interval corrected by the Fridericia Correction Formula values of >470msec; patient who is known to have congenital prolonged QT syndromes; or patient who is on medication known to cause prolonged QT interval on ECG.
11. Patient had received a transfusion (platelets or red blood cells) or colony-stimulating factors (e.g., granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) within 4 weeks before the exercise initiation.
12. Patient has underlying chronic lung disease, chronic obstructive pulmonary disease, metastatic lung disease, pleural effusions or pneumonitis.
13. Extensive non-oncological bone disease or presence of long-bones metastases or other symptomatic bone metastatic disease.
14. Significant peripheral sensory or motor neuropathy that could interfere with exercise program at investigator discretion.
15. Patient who are pregnant, breastfeeding, or expecting to conceive children during program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility (adherence) of a supervised physical exercise program in ovarian cancer patients on PARPi treatment. | 12 weeks
  Adherence to the program will be evaluated considering the total program completed/total program. Adherence per patient will be considered adequate if 70% of the planned program is exceeded. The percentage of patients who have been adherent to the program will be evaluated. Feasibility will be evaluated according to the percentage of adherent patients. The intervention will be considered feasible if the percentage of adherent patients is greater than or equal to 2/3 (66.6%) of the patients who give their consent to participate in the program and attend at least the first session.

SECONDARY OUTCOMES:
To evaluate the safety of a supervised physical exercise program in ovarian cancer patients on PARPi treatment. | 12 weeks
  Frequency of AEs occurring during the study, globally and program related will be described. Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
To assess fatigue levels at the end of intervention compared to levels prior to the start of the physical exercise program (Functional Assessment of Chronic Illness Therapy (FACIT-Fatigue questionnaire)). | 12 weeks
  Difference in fatigue levels at the end of intervention compared to levels prior to the start of the physical exercise and nutrition program (FACIT-Fatigue questionnaire). Score range: 0-52. Higher scores mean a better outcome.
To assess quality of life at the end of intervention compared to levels prior to the start of the physical exercise program european organization for research and treatment of cancer quality of life questionnaire core-30 (EORTC QLQ-C30). | 12 weeks
  Difference in quality of life at the end of intervention compared to levels prior to the start of the physical exercise and nutrition program (EORTC QLQ-C30). Score range: 0-100. A high score for the global health status represents a high quality of life.
To assess quality of life at the end of intervention compared to levels prior to the start of the physical exercise program european organization for research and treatment of cancer quality of life questionnaire ovarian 28 (EORTC QLQ-OV28). | 12 weeks
  Difference in quality of life at the end of intervention compared to levels prior to the start of the physical exercise and nutrition program (EORTC QLQ-OV28).
To assess quality of life at the end of intervention compared to levels prior to the start of the physical exercise program (PRO-CTCAE questionnaires). | 12 weeks
  Difference in quality of life at the end of intervention compared to levels prior to the start of the physical exercise and nutrition program (PRO-CTCAE questionnaires).
To compare biological data at the end of intervention compared to baseline data: baseline physical exercise level | 12 weeks
  Difference in biological data at the end of intervention compared to baseline data: physical exercise level (6 minute-walk test)
To compare fitness data at the end of intervention compared to baseline data: baseline physical exercise level | 12 weeks
  Difference in fitness data at the end of intervention compared to baseline data: physical exercise level (6 minute-walk test)
To compare biological data at the end of intervention compared to baseline data: baseline physical exercise level | 12 weeks
  Difference in biological data at the end of intervention compared to baseline data: physical exercise level International Physical Activity Questionnaire (IPAQ questionnaire).
To compare fitness data at the end of intervention compared to baseline data: baseline physical exercise level | 12 weeks
  Difference in fitness data at the end of intervention compared to baseline data: physical exercise level International Physical Activity Questionnaire (IPAQ questionnaire).
To compare biological data at the end of intervention compared to baseline data: baseline body composition | 12 weeks
  Difference in biological data at the end of intervention compared to baseline data: physical exercise level (body composition).
To compare fitness data at the end of intervention compared to baseline data: baseline body composition | 12 weeks
  Difference in fitness data at the end of intervention compared to baseline data: physical exercise level (body composition).
To compare biological data at the end of intervention compared to baseline data: baseline anthropometric values | 12 weeks
  Difference in biological data at the end of intervention compared to baseline data: physical exercise level (anthropometric values).
To compare fitness data at the end of intervention compared to baseline data: baseline anthropometric values | 12 weeks
  Difference in fitness data at the end of intervention compared to baseline data: physical exercise level (anthropometric values).
To compare biological data at the end of intervention compared to baseline data: baseline upper body strength/lower body strengt | 12 weeks
  Difference in biological data at the end of intervention compared to baseline data: physical exercise level (upper body strength (handgrip)/lower body strength (30 second sit to stand).
To compare fitness data at the end of intervention compared to baseline data: baseline upper body strength/lower body strengt | 12 weeks
  Difference in fitness data at the end of intervention compared to baseline data: physical exercise level (upper body strength (handgrip)/lower body strength (30 second sit to stand).
To compare psychological parameters at the end of intervention compared to baseline parameters:insomnia (ISI). | 12 weeks
  Difference in psychological parameters at the end of intervention compared to baseline parameters: Insomnia Severity Index (ISI).
To compare psychological parameters at the end of intervention compared to baseline parameters: depression and anxiety (HADS). | 12 weeks
  Difference in psychological parameters at the end of intervention compared to baseline parameters: Hospital Anxiety and Depression Scale (HADS).
To compare fatigue levels at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in fatigue levels at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare quality of life at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in quality of life at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare biological data at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in biological data at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare physical exercise level at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in physical exercise level at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare body composition at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in body composition at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare anthropometric values at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in anthropometric values at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare upper body strength (handgrip)/lower body strength parameters at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program. | 6 months
  Difference in upper body strength /lower body strength at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.
To compare psychological parameters at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program | 6 months
  Difference in psychological parameters at 3 months follow-up after the intervention vs levels prior to the start of the physical exercise program.

OTHER OUTCOMES:
To study and characterize different cell populations to evaluate the potential effect of physical exercise on immunosurveillance. | 12 weeks
  Difference in cell populations at the end the intervention compared to levels prior to the start of the physical exercise and nutrition program
To study and characterize different proteins to evaluate the potential effect of physical exercise on immunosurveillance. | 12 weeks
  Difference in proteins at the end the intervention compared to levels prior to the start of the physical exercise and nutrition program

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Cortés, MD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (4):
- Spain (4):
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid